CLINICAL TRIAL: NCT04534322
Title: An Expanded Access Program Protocol for Melphalan Flufenamide in Combination With Dexamethasone in Patients With Triple Class Refractory Multiple Myeloma
Brief Title: Expanded Access Program for Melphalan Flufenamide (Melflufen) in Triple Class Refractory Multiple Myeloma
Acronym: sEAPort
Status: Approved for marketing | Type: Expanded Access
Sponsor: Oncopeptides AB (Industry)
Responsible Party: Sponsor
Other Study IDs: OP-110
Record Dates: First submitted 2020-08-26; First posted 2020-09-01 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Relapsed and/or Refractory Multiple Myeloma
MeSH Terms: interventions — L-melphalanyl-p-L-fluorophenylalanine ethyl ester; melflufen; Dexamethasone

STUDY DESIGN:
Expanded Access Types: Intermediate, Treatment

INTERVENTIONS:
Drug: Melphalan Flufenamide — Melphalan flufenamide (melflufen) is an investigational peptide-drug conjugate (PDC) that targets aminopeptidases and rapidly releases alkylating agents into tumor cells.
  Other Names: melflufen
Drug: Dexamethasone — Dexamethasone, a synthetic adrenocortical steroid, is a white to practically white, odorless, crystalline powder. It is stable in air. It is practically insoluble in water.

SUMMARY:
To provide early treatment access and evaluate the safety of melflufen and dexamethasone in patients with triple class refractory (TCR) multiple myeloma (MM).

DETAILED DESCRIPTION:
This is a multicenter, expanded access program protocol to provide access to melflufen for patients with RRMM in medical need, who have progressive disease after they received a minimum of at least two prior lines of therapy, are triple-class refractory to at least one PI, at least one IMiD and at least one anti-CD38 mAb or intolerant to a specific therapeutic drug class. Patients with primary refractory MM are eligible to participate as long as they meet the criteria of being triple class refractory. They may meet these criteria for triple class refractory MM if they have received at least one PI, at least one IMiD, and at least one Anti-CD38 mAb in their first line treatment or have had at least 2 prior lines of therapy.

ELIGIBILITY:
Inclusion Criteria:

1. A clinically confirmed prior diagnosis of multiple myeloma with documented disease progression.
2. Triple-class refractory multiple myeloma (TCR MM). Triple-class refractory defined as refractory to at least one PI, at least one IMiD, and at least one Anti-CD38 mAb. Patients (with non-primary refractory MM) are required to have a minimum of at least 2 prior lines of therapy.

   Patients with primary refractory MM are eligible if they meet the criteria for TCR MM. They may meet these criteria for TCR MM if they have received at least one PI, at least one IMiD, and at least one Anti-CD38 mAb in their first line treatment or have had at least 2 prior lines of therapy.
3. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
4. Adequate organ function with the following laboratory results during screening (within 21 days) and immediately before treatment administration on Cycle1 Day1:

   * Absolute neutrophil count (ANC) ≥ 1,000 cells/mm3
   * Platelet count ≥ 75,000 cells/mm3 (75 x 109/L)
   * Hemoglobin ≥ 8.0 g /dL (Red blood cell (RBC) transfusions are permitted)
   * Total Bilirubin ≤ 1.5 x upper limit of normal (ULN), except patients diagnosed with Gilbert's syndrome AST (SGOT) and ALT (SGPT) ≤ 3.0 x ULN
   * Renal function: Estimated glomerular filtration rate (eGFR) by CKD-EPI formula of ≥ 45 mL/min.
5. Has not been enrolled in another melflufen clinical study and is not eligible for or does not have access to enroll in another ongoing clinical study of melflufen;
6. Contraception:

   1. Male patients: Agree to use contraception during the treatment period and for at least 3 months after the last dose of treatment and refrain from donating sperm during this period.
   2. Female patients: Eligible to participate if not pregnant or not breastfeeding, and at least one of the following conditions applies:

      * Not a woman of childbearing potential (WOCBP) or
      * A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 3 months after the last dose of treatment.

Exclusion Criteria:

1. Known platelet transfusion refractory (i.e. platelet count fails to increase by > 10,000 cells/mm3 after a transfusion of an appropriate dose of platelets);
2. Other malignancy diagnosed or requiring treatment within the past 3 years except for adequately treated basal cell carcinoma, squamous cell skin cancer, carcinoma in-situ of the cervix or breast, and very low and low risk prostate cancer patients in active surveillance.
3. Concurrent known or suspected (symptomatic) amyloidosis or plasma cell leukemia.
4. Any of the following treatments, within the specified timeframe:

   * Previous cytotoxic therapies, including cytotoxic investigational agents, for multiple myeloma within 3 weeks (6 weeks for nitrosoureas) prior to initiation of therapy.
   * IMiDs, PIs and or corticosteroids within 2 weeks prior to initiation of therapy.
   * Other investigational therapies within 4 weeks of initiation of therapy.
   * Prednisone up to but no more than 10 mg orally q.d. or its equivalent for symptom management of comorbid conditions is permitted but dose should be stable for at least 7 days prior to initiation of therapy.
5. Prior stem cell transplant (autologous and/or allogeneic) within 6 months of initiation of therapy.
6. Prior allogeneic stem cell transplant with active graft-versus-host- disease (GVHD);
7. Prior major surgical procedure or radiation therapy within 4 weeks of the first dose of treatment (this does not include limited course of radiation used for management of bone pain within 7 days of initiation of therapy);
8. Prior treatment with melflufen

Key eligibility criteria listed and is not all inclusive

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Highlands Oncology Group, Springdale, Arkansas
  - Beacon Cancer Care, Coeur d'Alene, Idaho
  - University of Illinois Cancer Center, Chicago, Illinois
  - Weill Cornell Medicine - Multiple Myeloma Center, New York, New York
  - Gabrail Cancer Center, Canton, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Prisma Health Cancer Institute, Greenville, South Carolina
  - Texas Oncology, Dallas, Texas
  - Community Cancer Trials of Utah, Ogden, Utah
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Northwest Medical Specialties, Tacoma, Washington